CLINICAL TRIAL: NCT04624490
Title: Hyperpolarized 129Xe MR Imaging of Lung Function in Healthy Volunteers and Subjects With Pulmonary Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Mario Castro, MD, MPH (Other)
Responsible Party: Sponsor-Investigator, Mario Castro, MD, MPH, Division Chief, Pulmonary, Critical Care and Sleep Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00146119
Record Dates: First submitted 2020-10-31; First posted 2020-11-10 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Asthma; COPD; Interstitial Lung Disease; Cystic Fibrosis; Pulmonary Hypertension; Pulmonary Infection; Other Lung Disease
Keywords: Hyperpolarized 129Xe MRI
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Lung Diseases, Interstitial; Cystic Fibrosis; Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hyperpolarized 129Xe (Experimental): Administration of hyperpolarized xenon during MRI (up to 1L doses) to develop imaging methods and assess pulmonary function in adults.
  Interventions: Drug: Hyperpolarized Xe129

INTERVENTIONS:
Drug: Hyperpolarized Xe129 — During MRI scanning, subject will inhale hyperpolarized xenon gas for a maximum of 16 seconds per scan, with a maximum of 4 MR scans + Calibration in a given imaging session.
  Other Names: HP Xenon

SUMMARY:
The purpose of this study is to develop and evaluate the usefulness of hyperpolarized (HP) 129Xe gas MRI for regional assessment of pulmonary function.

DETAILED DESCRIPTION:
This is an unblinded, open-label study with ~160 subjects with diagnosed pulmonary disease and ~100 healthy controls. Subjects to be enrolled will include males and females 18-80 years old. Evaluation will be on an outpatient basis. Imaging will be done on a single day and will involve administration of up to four 1-liter doses of HP 129Xe plus one 129Xe calibration dose (~300-400mL HP 129Xe). In addition to 129Xe MRI, a series of anatomical conventional 1H MR images will be collected including a localizer scan, breath-hold spin echo image, and breath-hold steady-state free precession image to highlight the vasculature. All subjects will be evaluated at one center: The University of Kansas Medical Center, KS USA.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Subject has no diagnosed pulmonary conditions
* Ability to read and understand English or Spanish

Subjects with Lung Disease:

* Subject has a diagnosis of pulmonary dysfunction made by a physician
* No acute worsening of pulmonary function in the past 30 days
* Ability to read and understand English or Spanish

Exclusion Criteria:

* MRI is contraindicated based on responses to MRI screening questionnaire
* Subject is pregnant or lactating
* Subject does not fit into 129Xe vest coil used for MRI
* Subject cannot hold his/her breath for 15-16 seconds
* Subject deemed unlikely to be able to comply with instructions during imaging
* Oxygen saturation <88% on room air or with supplemental oxygen
* Cognitive deficits that preclude ability to provide consent
* Institutionalization

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2020-11-02 (Actual); Primary Completion 2025-10-26 (Estimated); Study Completion 2026-10-26 (Estimated)

PRIMARY OUTCOMES:
RBC/Barrier Ratio | Day 1
  Ratio of xenon signal dissolved in RBCs to xenon signal dissolved in Barrier Tissues

SECONDARY OUTCOMES:
ADC | Day 1
  Apparent Diffusion Coefficient of Xenon Gas in the lungs
Ventilation Defect Percentage | Day 1
  Percentage of the Lungs with ventilation signal below a threshold level

CONTACTS AND LOCATIONS:
Overall Officials: Peter Niedbalski, PHD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States